CLINICAL TRIAL: NCT00617617
Title: The Specific Role of Isoflavones in Reducing Prostate Cancer Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Cognis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCC-12835; NCI #4031; CA 81920; NCT00027950 (obsolete NCT alias)
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2010-02

CONDITIONS: Prostate Cancer
Keywords: isoflavones; soy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Dietary Supplement: Prevastein HC®
  Interventions: Dietary Supplement: Prevastein HC®
- B (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Prevastein HC® — Experimental Group - Participants in the experimental group will consume an isoflavones supplement in the form of Prevastein HC®, which will deliver 80 mgs (40 mg/dose) biologically active isoflavones.
  Arms: A
Other: Placebo — Control Group - Control Group participants will receive an identical placebo.
  Arms: B

SUMMARY:
The purpose of this research study is to determine if giving men with early stage (Grade 1-2) prostate cancer dietary supplement from soybeans called isoflavones, will change their blood hormone levels. Isoflavones are substances found in a high concentration in soybeans that are converted in the intestines to hormone-like compounds which are similar to estrogen. They are also thought to have cancer fighting properties. Clinical trials suggest that isoflavones can increase certain sex hormones, which results in the slower production of prostate cancer cells. This study will determine if adding isoflavones (supplied as Prevastein HC®) 80 mg/day in a pill form can change your risk factors that cause early stage prostate cancer to progress to more advanced disease.

DETAILED DESCRIPTION:
To prevent biasing the outcome of the study, this is a double-blind study design, where both the trialists and the participants are blinded to the specific nature of the product (isoflavones and placebo). Participants in both groups will be discouraged from increasing their intake of dietary isoflavones in the form of tofu, soy beans, soy milk, etc. In addition, the intervention does not include active counseling on dietary modification and supplementation of any one group. Monthly appointments will be made for all participants for data collection and toxicity assessment.

Schema:

This is a controlled, randomized, double blinded clinical trial, having one experimental and one control group (n - 75/arm). Participants in the experimental group will consume an isoflavones supplement in the form of Prevastein HC®, which will deliver 80 mgs (40 mg/dose) biologically active isoflavones and those in the control group will receive an identical placebo. The isoflavones supplement and the placebo tablets will be manufactured and packaged by Cognis Corporation.

1. Isoflavones will be supplied at no charge by Cognis Corporation, LaGrange, Illinois as Prevastein HC®. Each Prevastein HC® tablet delivers 20 mg biologically active isoflavones, which is available for absorption. Participants will consume 2 tablets twice daily (with meals) in addition to their usual diet.
2. Placebo will be supplied at no charge by Cognis Corporation, LaGrange, Illinois as an indistinguishable tablet. Participants will consume 2 tablets twice daily (with meals) in addition to their usual diet.
3. A standardized multivitamin will be supplied at no charge.

ELIGIBILITY:
Inclusion Criteria:

* Males, between the ages of 50 and 80
* Diagnosed with grade 1-2 prostate cancer (Gleason Score 2 to 6) Note: patients with a Gleason primary pattern 4 (4+1 or 4+2) are not eligible.
* No prior or current therapy for prostate cancer
* No other history of cancer except non-melanoma skin cancer
* No known history of hepatic and/or renal disease
* No evidence of prostatitis or urinary tract infection (men being treated with antibiotics may be enrolled 30 days after completion of therapy given that they still meet all other eligibility criteria)
* No antibiotic use within 30 days of registration
* Close to ideal body weight(Body Mass Index no greater than 32 Kg/m²)
* Omnivorous diet
* Able and willing to give written consent

Exclusion Criteria:

* Less than 50 years or over 80 years of age
* Prostate cancer beyond grade 2 (Gleason Score greater than 6)
* Gleason primary pattern 4 (4+1 or 4+2)
* Prior or planned treatment for prostate cancer of any stage
* Prior history of other cancer except non-melanoma skin cancer
* Current use of nutritional supplements, including modular supplements of other agents with antioxidant properties e.g. retinoids, beta-carotene, and isoflavones
* Allergy to study agent
* Known history of hepatic or renal disease
* Body Mass Index greater than 32 Kg/m²
* Vegetarian/vegan diet
* Diet high in soy products (men who routinely consume a diet high in soy products may be enrolled 30 days after eliminating soy product from the diet)
* Prostatitis or urinary tract infection
* Treatment with antibiotics within 30 days of registration

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2002-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Observe the effects of the 12 - week intervention with isoflavones on sex hormones and PSA, a marker of disease progression. | 12 week treatments

CONTACTS AND LOCATIONS:
Overall Officials: Nagi B. Kumar, PhD., RD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States